CLINICAL TRIAL: NCT01734109
Title: A 12-week, Single Site, Randomized Controlled Trial to Compare the Efficacy of Quantum NPWT With and Without Simultaneous Irrigation Versus Standard of Care on Reduction of the Volume of Stage III/IV Pressure Ulcers.
Brief Title: Efficacy of Quantum NPWT With Simultaneous Irrigation on Reduction of Wound Volume in Stage III/IV Pressure Ulcers.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Innovative Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITIQ002A
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Pressure Ulcers
Keywords: Negative Pressure Wound Therapy; Irrigation Therapy; Pressure Ulcers; Sacral Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care - Wound Care (Placebo Comparator): Standard, acceptable local wound care management, consisting of topical treatments, chemical debriders, or light bedside debridement.
- Quantum NPWT (Active Comparator): Intervention with Quantum NPWT to Standard III/IV pressure ulcers for 12 weeks.
  Interventions: Device: Quantum Negative Pressure Wound Therapy Device
- Quantum NPWT with Irrigation (Active Comparator): NPWT with the Quantum device, with the addition of simultaneous irrigation using 0.25% acetic acid.
  Interventions: Device: Quantum Negative Pressure Wound Therapy Device

INTERVENTIONS:
Device: Quantum Negative Pressure Wound Therapy Device — To compare the additional benefit of Quantum Negative pressure wound therapy device with and without simultaneous irrigation.
  Other Names: Quantum NPWT
  Arms: Quantum NPWT; Quantum NPWT with Irrigation

SUMMARY:
Negative-pressure wound therapy (NPWT) is an important adjunct for management of wounds, and promotes granulation tissue and angiogenesis. Despite these known means for facilitation of wound management, further research is needed to examine whether this modality is superior to other currently used options, thus defining clear indications for and benefits of NPWT. This would also help establish the role of combination therapy, using NPWT with simultaneous irrigation or other forms of dressings. This study aims to compare treatment efficacy of NPWT, NPWT plus proprietary simultaneous irrigation, and traditional hospital standard of care for treatment of grade III & IV pressure ulcers. Primary endpoint of this study is comparison of reduction of wound volume between the three treatment arms; and secondary endpoints include bacterial load, rate of wound healing, preparation for grafting, and pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between the ages of 18 and 70
* Any patient with a stage III/IV pressure ulcer of the size large enough to indicate use of Negative Pressure Treatment.

Exclusion Criteria:

* Clinical evidence of active, gross infection.
* Patient or patient's guardian refuses consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-09 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of reduction in wound volume between Quantum with Irrigation v Standard of Care | 12-weeks
  Comparison of reduction in wound volume between Quantum with Irrigation versus standard of care over 12 weeks treatment period.

SECONDARY OUTCOMES:
Comparison of reduction in wound volume between Quantum with Irrigation v Quantum without irrigation | 12 weeks
  Comparison of reduction in wound volume between Quantum with Irrigation versus Quantum without irrigation over 12 weeks measurement period.

OTHER OUTCOMES:
Pain | 12 weeks
  Weekly assessment of pain using standard VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J Berriman, Ph.D., Study Director — Innovative Therapies, Inc.; Kenneth Moquin, MD, Principal Investigator — Henry Ford Hospital System
Locations (1):
- Henry Ford Hospital System, Detroit, Michigan, United States